CLINICAL TRIAL: NCT05731869
Title: Investigation of the Effect of Epicondylitis Band and Wrist Orthosis on Extensor Muscle Activity and Upper Extremity Functions
Brief Title: Investigation of the Effect of Epicondylitis Band and Wrist Orthosis
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/058
Record Dates: First submitted 2023-02-09; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Splints
Keywords: surface electromyography; muscle activation; orthosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: The group measured without the use of orthoses and tapes
- Epicondylitis Band Group: Group measured with epicondylitis band
  Interventions: Other: epicondylitis band
- Wrist Orthosis Group: Group measured with wrist orthosis
  Interventions: Other: wrist orhosis

INTERVENTIONS:
Other: epicondylitis band — An off-the-shelf lateral epicondylitis tape in S-M-L dimensions was used distal to the lateral epicondylitis.
  Groups: Epicondylitis Band Group
Other: wrist orhosis — Wrist orthosis of the shelf was used in sizes S-M-L, covering the hand and wrist.
  Groups: Wrist Orthosis Group

SUMMARY:
Muscles that are frequently injured in the extensor group are extensor carpi radialis longus, extensor carpi radialis brevis, and extensor digitorum communis. Injury of these muscles is seen as lateral epicondylitis in the clinic. Physiotherapy techniques are frequently applied in the management of diseases related to forearm extensor muscles such as lateral epicondylitis. Various orthoses such as lateral epicondylitis band, wrist orthosis, dynamic extensor brace are used for this. Studies have been conducted on pain, hand function and orthosis satisfaction of different types of lateral epicondylitis orthoses, and the number of studies investigating the effects on muscle activation is insufficient.Therefore, the aim of the study is to examine the effects of different types of orthoses used for the forearm extensor group on extensor muscle activation and upper limb functions.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-45 years old
* Right upper extremity dominant
* No upper extremity limitation in activities of daily living
* Volunteer individuals

Exclusion Criteria:

* With orthopedic, neurological and rheumatological problems in the upper extremity
* Entrapment neuropathy, TOS, cervical radiculopathy, and cervical disc herniation
* History of upper extremity injury or surgery in the last 6 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
muscle activation | one hour
  A superficial EMG system will be used to measure signals from the extensor carpi radialis longus/brevis and extensor carpi digitorum communis muscles.Electrodes will be placed according to SENIAM criteria.The signals received from the muscles of the individuals will be recorded during grasping. As a result, the average muscle activations of the muscles during the activity will be numerically recorded in %MVIC.

SECONDARY OUTCOMES:
hand function | one hour
  Jebson Taylor Hand Function Test, which includes daily life activities (writing, eating, etc.) and consists of 7 sub-parameters, was applied to measure hand function. The score is recorded in seconds and the score gets worse as the second increases.
satisfaction level | one hour
  The OPUS questionnaire was used to measure the participants' orthotic satisfaction. The OPUS questionnaire evaluates the weight, durability, aesthetics, ease of putting on, skin and clothing problems, comfort, and the pain-reducing effect of the orthosis associated with the orthosis. The higher the score, the higher the level of satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Mustafa Sarı, Çankaya, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Sari M, Ozturk D, Bek N. Comparison of two different orthoses used in the treatment of lateral epicondylitis. Prosthet Orthot Int. 2025 Feb 1;49(1):127-132. doi: 10.1097/PXR.0000000000000345. Epub 2024 Mar 22. PMID 38517366